CLINICAL TRIAL: NCT02985554
Title: Phase I Study to Assess the Tolerability and Efficacy of Nivolumab as Single Agent to Eliminate Minimal Residual Disease and Maintain Remission in Patients With Hematologic Malignancies After Allogeneic Stem Cell Transplantation
Brief Title: Phase I Study to Assess the Tolerability and Efficacy of Nivolumab in Patients With Hematologic Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study stopped early due to slow accrual and safety concerns.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB16-0888
Record Dates: First submitted 2016-12-01; First posted 2016-12-07 (Estimated); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Hematologic Malignancies
Keywords: hematologic malignancies; allogeneic stem cell transplantation (allo-SCT)
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): Nivolumab will be administrated intravenously. Standard dose escalation will be used for the intensification phase with starting dose at 1m/kg every 2 weeks for 4 doses.
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab dose escalation will be used for the intensification phase with starting dose at 1m/kg every 2 weeks for 4 doses.
  Other Names: Opdivo

SUMMARY:
This is an open-label, dose escalation Phase I study to evaluate the tolerability and efficacy of single agent of Nivolumab as maintenance treatment to prevent relapse in patients with hematologic malignancies after allogeneic stem cell transplantation. Approximately 29 patients will be enrolled, where about 6-12 patients will be included on the dose escalation phase and 20 patients will be on the expansion cohort at maximal tolerated dose.

DETAILED DESCRIPTION:
Nivolumab will be administrated intravenously. Standard dose escalation will be used for the intensification phase with starting dose at 1m/kg every 2 weeks for 4 doses. The DLT observation period is 29 days starting with the first dose taken on Day 1, The study treatment will continue until one of the discontinuation criteria is met. Each dose level (1-2) will be tested using the 3+3 design. If level 2 of 3mg/kg is reached without DLTs, 3mg/kg will be used for the dose expansion cohort. After the intensification phase, patients will start Nivolumab every 12 weeks maintenance phase till 2 years post allo-SCT. Patients will also receive best supportive care (BSC), including blood product transfusions, antimicrobials, and (as appropriate) granulocyte colony stimulating factors for neutropenic infection or poor graft function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hematologic malignancies status post allogeneic SCT without evidence of disease relapse, active GVHD or history of more than Stage I skin acute GVHD; and off immunosuppression for at least 4 weeks. At least 60 days after allo-SCT.
* Patients with high risk myeloid or lymphoid malignancies at stem cell transplant following ASBMT criteria (http://www.asbmt.org/displaycommon.cfm?an=1&subarticlenbr=35, under disease classification), including but not limited to conditions listed. Refractory acute myelogenous or lymphoid leukemia Relapsed acute myelogenous or lymphoid leukemia Myelodysplastic syndromes with 5% or more blasts Chronic myelogenous leukemia in chronic phase 3 or more, blast phase presently, or second accelerated phase, Recurrent or refractory malignant lymphoma or Hodgkin's disease with less than a partial response at transplant High risk chronic lymphocytic leukemia defined as no response or stable disease to the most recent treatment regimen.
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of nivolumab in patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* ECOG/Karnofsky performance status of 0 or 1 (Karnofsky ≥70%, see Appendix A).
* Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to treatment.
* leukocytes ≥2000/mcL
* absolute neutrophil count ≥1,000/mcL(In the absence of growth factor support)
* platelets ≥50,000/mcL or recovery to the baseline count(in the absence of transfusion)Hgb >9.0g/dL
* total bilirubin ≤1.5× institutional upper limit of normal (ULN) (except patients with Gilbert Syndrome, who can have total bilirubin <3.0 mg/dL)
* AST(SGOT)/ALT(SGPT) ≤3 × ULN 17
* Serum creatinine ≤1.5× ULN OR
* creatinine clearance (CrCl) ≥40 mL/min (if using the Cockcroft-Gault formula below): Female CrCl = (140 - age in years) x weight in kg x 0.85 72 x serum creatinine in mg/dL Male CrCl = (140 - age in years) x weight in kg x 1.00 72 x serum creatinine in mg/dL
* The effects of nivolumab on the developing human fetus are unknown. For this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. WOCBP should use an adequate method to avoid pregnancy for 23 weeks) after the last dose of investigational drug Nivolumab. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of nivolumab. Women must not be breastfeeding. Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception. Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational product. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product. These durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately. 18
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* History of allergy to study drug components.
* Patients who have disease relapse, active GVHD or history of more than Stage 1 skin acute GVHD, history of cGVHD.
* Patients with active infection, un-resolving more than grade 2 transplant-related toxicities.
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (AEs) due to agents administered more than 4 weeks earlier.
* Patients who are receiving any other investigational agents.
* Patients with known CNS involvement may be excluded because of poor prognosis and concerns regarding progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. However, if CNS disease is cleared before the treatment with Nivolumab, patients could be allowed if no permanent CNS damage.
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because Nivolumab is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Nivolumab, breastfeeding should be discontinued if the mother is treated with Nivolumab.
* Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) might be enrolled if the viral load by PCR is undetectable with/without active treatment and absolute lymphocyte count >= 350/ul. Patients with a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection might be enrolled if the viral load by PCR is undetectable with/without active treatment.
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as SLE, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease. Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible. Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intraarticular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).

Physiologic replacement doses of systemic corticosteroids are permitted, even if <10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.

* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study.eligible. Patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible.
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event).
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease. Patients are permitted to use topical, ocular, intraarticular, intranasal, and inhalational corticosteroids (with minimal systemic absorption).

Physiologic replacement doses of systemic corticosteroids are permitted, even if <10 mg/day prednisone equivalents. A brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted.

* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, GI obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of Nivolumab | 24 months
  The maximum tolerated dose (MTD) of Nivolumab in patients with hematologic malignancies after allo-SCT.

SECONDARY OUTCOMES:
Number of type of adverse events | 24 months
  To evaluate the toxicities of Nivolumab as maintenance treatment after allogeneic stem cell transplantation (allo-SCT).
Incidence of non-relapse mortality | From the date of therapy to the date of non-relapse death, whichever came first, assessed up to 100 months
Time until progression free survival | From start date of therapy to the first documented disease relapse or death from any cause, whichever may come first, assessed up to 100 months
Time until overall survival | From start date of therapy to death from any cause, whichever may come first, assessed up to 100 months

OTHER OUTCOMES:
Differences in pre- and post treatment levels of T cell subsets and T cell activation status | 24 months
  To perform an exploratory analysis on the frequencies, absolute numbers and subsets of T cells (including regulatory T cells) in Nivolumab treated patients.
Differences in pre- and post treatment levels for inspection of changes in "clonality" of T cell repertoire between blood samples | 24 months
  To perform deep sequencing of TCR-alpha and TCR-beta chains on polyclonal T cells at baseline and at subsequent time points during nivolumab treatment. Changes in levels of responders versus nonresponders will be analyzed using a non-parametric Wilcoxon rank-sum test.
Quantitative RT-PCR (qPCR) results in peripheral blood and bone marrow samples | 24 months
  To monitor MRD by WT1 PCR during Nivolumab treatment in AML/MDS patients. The differences will be assessed using a conventional T-test or Wilcoxon rank-sum test.

CONTACTS AND LOCATIONS:
Overall Officials: Hongtao Liu, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States